CLINICAL TRIAL: NCT02336464
Title: Impact of DYSpnea on the ouTcome of Patients Admitted for an Acute RESpiratory Failure in the intenSive Care Unit
Brief Title: Impact of Dyspnea on Patients in the Intensive Care Unit
Acronym: DYSTRESS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K120103
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2018-05

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although pain has been extensively studied in ICU patients, only a few studies have focused on dyspnea, which is experienced by 50% of mechanically ventilated patients. The purpose of the present study is to determine whether dyspnea in intensive care unit patients is associated with a higher length of stay in the ICU and a higher incidence of post traumatic stress disorders.

DETAILED DESCRIPTION:
Intensive care unit (ICU) patients are continuously exposed to various unpleasant sensations that are as many sources of discomfort. If, growing attention has been given to the detection and treatment of pain, very little attention has been given to dyspnea. However, there is growing evidence suggesting that dyspnea is frequent and severe in mechanically ventilated ICU patients. In mechanically ventilated ICU patients, dyspnea is independently associated with anxiety and mechanical ventilation itself. Indeed, an optimization of ventilator settings alleviates dyspnea in 35% of patients.

Various arguments suggest that dyspnea contributes to the dark experience of ICU and participates to the genesis of post traumatic stress disorders. In addition, dyspnea is associated with a longer duration of mechanical ventilation.

Large multicentre studies are however lacking. The aims of the present multicentre study are 1) to quantify the prevalence of dyspnea in a large population of ICU mechanically ventilated patients, 2) to examine the link between the level of dyspnea and the occurrence of adverse events in the ICU, 3) to determine whether dyspnea in intensive care unit patients is associated with a higher length of stay in the ICU and a higher incidence of post traumatic stress disorder associated symptoms.

ELIGIBILITY:
Inclusion criteria:

* Invasive mechanical ventilation in the ICU for > 24 hours
* Remaining stay in the ICU estimated > 24 hours

Exclusion criteria :

* RASS <-2 or >+2
* Delirium (defined according to CAM-ICU)
* Severe cognitive impairment or severe psychiatric disease
* Patient who does not understand French
* Severe depthless
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aims of the present multicentre study are 1) to quantify the prevalence of dyspnea in a large population of ICU mechanically ventilated patients, 2) to examine the link between the level of dyspnea and the occurrence of adverse events in the ICU, 3) to determine whether dyspnea in intensive care unit patients is associated with a higher length of stay in the ICU and a higher incidence of post traumatic stress disorder associated symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04-13 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | 3 months
incidence of post traumatic stress disorders | 3 months

SECONDARY OUTCOMES:
Anxiety and depression (Hamilton anxiety and depression scale) | 3 months
  Hamilton anxiety and depression scale
Quality of life (Short-Form 36) | 3 months
  Short-Form 36
Pain (Visual Analogic Scale) | 3 months
  Visual Analogic Scale
Quality of Sleep (Pittsburgh Scale) | 3 months
  Pittsburgh Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alesxandre Demoule, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demoule A, Hajage D, Messika J, Jaber S, Diallo H, Coutrot M, Kouatchet A, Azoulay E, Fartoukh M, Hraiech S, Beuret P, Darmon M, Decavele M, Ricard JD, Chanques G, Mercat A, Schmidt M, Similowski T; REVA Network (Research Network in Mechanical Ventilation). Prevalence, Intensity, and Clinical Impact of Dyspnea in Critically Ill Patients Receiving Invasive Ventilation. Am J Respir Crit Care Med. 2022 Apr 15;205(8):917-926. doi: 10.1164/rccm.202108-1857OC. PMID 35061577